CLINICAL TRIAL: NCT02921477
Title: Open Label Study for the Use of Tyrosine Kinase Inhibitors for Treatment of Cognitive Decline Due to Degenerative Dementias
Brief Title: Study for the Use of TKIs for Treatment of Cognitive Decline Due to Degenerative Dementias
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Neurological Associates of West Los Angeles (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Sheldon Jordan, Neurologist, Neurological Associates of West Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 062016
Record Dates: First submitted 2016-09-28; First posted 2016-10-03 (Estimated); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Mild Cognitive Impairment; Dementia
Keywords: tyrosine kinase inhibitor; bosutinib; bosulif
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bosutinib Treatment Arm (Experimental): Subjects will be administered the initial dose of bosutinib, with dosage progressively increased over the course of the study. The initial dose of bosutinib is 100 mg tablet, once per day. The dose will be increased as tolerated up to 300 mg per day. The dose will be increased by 100 mg each month if the lower dose is tolerated without significant side effects. That is to say, the subject will take 100 mg/day every day for the first month, 200 mg/day every day for the second month, and 300 mg/day every day for the third month and for the remainder of the study, provided that adverse reactions do not prohibit continuation at this dosage. Stopping and dose reduction rules for reported adverse reactions have been taken from the package insert of bosutinib. The duration of treatment is 1 year.
  Interventions: Drug: bosutinib

INTERVENTIONS:
Drug: bosutinib
  Other Names: bosulif; TKI

SUMMARY:
The present study is designed as an open label study of patients with mild cognitive impairment or dementia to evaluate longer term tolerability and potential efficacy of tyrosine kinase inhibitors. Baseline and outcome measures in this study utilize validated tests that are appropriate for repeated measures which are not affected by practice effects. Advantages of this study include the fact that the neuropsychological testing instruments and advanced MRI imaging protocols that have been in routine clinical deployment provide for a high degree of availability and reliability for diagnosis and for monitoring change of status. Quality assurance is tightly controlled. The study population is sufficiently broad and the conditions of interest are sufficiently prevalent so that recruitment of the projected numbers of subjects is not a limiting factor.

For a Phase I trial there is a proposed 150 patient sample to determine the frequency of common side effects in the population that is being studied. Subjects will be administered the initial dose of bosutinib, with dosage progressively increased over the course of the study. The initial dose of bosutinib is 100 mg tablet, once per day. The dose will be increased as tolerated up to 300 mg per day.

All subjects will be started at 100 mg/day and the dose will be increased by 100 mg each month if the lower dose is tolerated without significant side effects. That is to say, the subject will take 100 mg/day every day for the first month, 200 mg/day every day for the second month, and 300 mg/day every day for the third month and for the remainder of the study, provided that adverse reactions do not prohibit continuation at this dosage. The investigators will be using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 to monitor, evaluate, and report adverse reactions on an ongoing basis. Stopping and dose reduction rules for reported adverse reactions have been taken from the package insert of bosutinib.

DETAILED DESCRIPTION:
In order for a subject to be considered for this study, the following criterion is required:

• Cognitive decline with mild cognitive impairment (Clinical Dementia Rating Stage 0.5) through moderate dementia (CDR Stages 1 and 2)

All patients, according to routine best practices will have an evaluation including neurological interview and examination to screen for reversible causes of cognitive change such as depression, substance abuse, vitamin deficiency and systemic illness. All patients will have a Beck Depression scale and blood tests for B12 and thyroid hormone. Patients will have an EKG, in particular to screen for QT prolongation which is a relative counterindication for use of tyrosine kinase inhibitor therapy.

According to the package insert for bosutinib, the investigators are proposing to use an age range and dosage route that is comparable and overlapping with routine application of this drug. In addition, the investigators are proposing dosage ranges that are substantially lower than usually recommended for treatment of leukemia.

The QDRS scale will be given to all patients; a cut off score of 1.5 has been used qualify patients with a dementia score (CDR) of 0.5 (ref 19).

All patients will have a lumbar puncture for ABeta 42 and Tau proteins for Alzheimer's Spectrum. This spinal fluid examination has been shown to be both sensitive and specific for Alzheimer's disease (ref 20). Cerebrospinal fluid (CSF) tau levels are also elevated in alpha synucleinopathy and frontotemporal lobar degeneration (ref 21). The lumbar puncture is performed once at entry.

All patients will have an advanced MRI of the brain to include volume measurement of the hippocampus (ref 22), arterial spin labeling (ASL) perfusion scan (ref 23) and MRS of prefrontal, precuneus, hippocampus and occipital lobe. Patients with cognitive decline have decreased perfusion in temporal parietal or frontal regions of the brain with ASL perfusion, or show characteristic change in MRS or volumetric evaluation compared to aged matched control subjects. MRI will also demonstrate if patients have tumors, hydrocephalus, subdural hematomas and other structural etiologies of cognitive decline.

On entry, patients will have CDR stage of at least 0.5 and at least one abnormal imaging biomarker and none of the exclusion criteria below. Baseline, six months, twelve months, eighteen months and two year (completion) testing will include the Quick Dementia Rating System (QDRS) for staging and the following battery of tests:

* the Repeatable Battery for Assessment of Neuropsychological Status (RBANS),
* Standardized 25 foot timed gait test
* the Nine Hole Pegboard Test,
* Montreal Cognitive Assessment Test versions 1,2,3 (MOCA),
* Brain imaging will be repeated at one year and two years. CSF studies have demonstrated good sensitivity and specificity for mild cognitive impairment (MCI) and dementia of the Alzheimer's type (ref 5). MRI volumetrics, perfusion scans and magnetic resonance spectroscopy (MRS) have shown to be of excellent discriminating value among Alzheimer's dementia (AD), Parkinson's spectrum degeneration (PDD/DLB) and frontal temporal lobar degeneration (FTLD) subgroups and is responsive to change as patient's progress from MCI to dementia (ref 6).

The rationale behind this criterion is supported by the importance that the subject is cognitively able to effectively speak, listen, and read in English, and has the cognitive capacity to give informed consent.

All subjects will be started at 100 mg/day and the dose will be increased by 100 mg each month if the lower dose is tolerated without significant side effects. Adverse reactions will be scaled according to the CTCAE v.5. If the subject experiences severe adverse reactions at any dose, or if the subject requires dose reduction for toxicity from a dose of 100 mg/day, the subject will be removed from the study. If the subject experiences moderate adverse reactions at a dose >100 mg/day, the dose will be reduced by 100 mg and maintained at the lower dose for 1 month. If the subject experiences moderate or severe adverse reactions at this lower dose, the subject will be removed from the study. After 1 month, the dose will again be increased by 100 mg. If the subject does not experience any adverse reactions at this elevated dose, he/she will resume with the original up-titration schedule (i.e. increase by 100 mg every month up to 300 mg/day). If the subject experiences moderate symptoms at this elevated dose, the dose will again be reduced by 100 mg and will be maintained at this lower dose as the maximally tolerated dose.

The duration of treatment is 1 year. To minimize risk, subjects will be seen regularly for toxicity monitoring during the first month of treatment, and biweekly during the second month of treatment. On weeks when the subject is not in for a visit, subject status will be assessed on the basis of phone calls with the respective care taker. The care taker will be determined during the QDRS staging at the time of the initial consultation. The care taker is an individual who is intimately familiar and in close contact with the subject. After the first two months, visits will be on a monthly basis. Mild, moderate, and severe adverse reactions will be reported on an ongoing basis. The rationale for such extended administration is to allow for a more reliable assessment of tolerability. The primary endpoint in evaluating tolerability will be how many of the initial 20 subjects are discontinued due to adverse reactions. Subjects will be discontinued if they have moderate or severe adverse reaction ratings according to the CTCAE, which are not remediable by dosage reduction.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive decline with mild cognitive impairment (Clinical Dementia Rating Stage 0.5) through moderate dementia (CDR Stages 1 and 2)

Exclusion Criteria:

* Subjects with a history of hypersensitivity to bosutinib
* Subjects with contraindications for lumbar puncture, such as bleeding abnormalities, use of anticoagulant medications, and local skin or spine abnormalities
* Reversible causes of cognitive impairment that explains the clinical status entirely, such as hypothyroidism, depression
* Advanced stages of any terminal illness or any active cancer that requires chemotherapy
* Pre-existing renal impairment
* Pre-existing hepatic impairment
* QT prolongation
* Significant cytopenia
* Cardiovascular, cerebrovascular, and peripheral vascular arterial thrombosis
* Women who are pregnant, may become pregnant, or are breastfeeding
* Women of child-bearing potential and male participants with female partners who are of child-bearing potential
* Subjects unable to give informed consent or in vulnerable categories, such as prisoners

Ages: 45 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients who are discontinued due to tolerability issues related to treatment | 1 year
  Outcome goal to determine safety and tolerability of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, MD, Principal Investigator — Neurological Associates of West Los Angeles
Locations (1):
- Neurological Associates of West LA, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carneiro BA, Kaplan JB, Giles FJ. Tyrosine kinase inhibitor therapy in chronic myeloid leukemia: update on key adverse events. Expert Rev Hematol. 2015 Aug;8(4):457-79. doi: 10.1586/17474086.2015.1041910. Epub 2015 May 4. PMID 25938861
- [Background] Hebron ML, Lonskaya I, Moussa CE. Nilotinib reverses loss of dopamine neurons and improves motor behavior via autophagic degradation of alpha-synuclein in Parkinson's disease models. Hum Mol Genet. 2013 Aug 15;22(16):3315-28. doi: 10.1093/hmg/ddt192. Epub 2013 May 10. PMID 23666528
- [Background] Lonskaya I, Hebron M, Chen W, Schachter J, Moussa C. Tau deletion impairs intracellular beta-amyloid-42 clearance and leads to more extracellular plaque deposition in gene transfer models. Mol Neurodegener. 2014 Nov 10;9:46. doi: 10.1186/1750-1326-9-46. PMID 25384392
- [Background] Tapiola T, Alafuzoff I, Herukka SK, Parkkinen L, Hartikainen P, Soininen H, Pirttila T. Cerebrospinal fluid beta-amyloid 42 and tau proteins as biomarkers of Alzheimer-type pathologic changes in the brain. Arch Neurol. 2009 Mar;66(3):382-9. doi: 10.1001/archneurol.2008.596. PMID 19273758
- [Background] Targosz-Gajniak MG, Siuda JS, Wicher MM, Banasik TJ, Bujak MA, Augusciak-Duma AM, Opala G. Magnetic resonance spectroscopy as a predictor of conversion of mild cognitive impairment to dementia. J Neurol Sci. 2013 Dec 15;335(1-2):58-63. doi: 10.1016/j.jns.2013.08.023. Epub 2013 Aug 27. PMID 24035276
- [Background] Hebron M, Moussa CE. Two sides of the same coin: tyrosine kinase inhibition in cancer and neurodegeneration. Neural Regen Res. 2015 Nov;10(11):1767-9. doi: 10.4103/1673-5374.165320. No abstract available. PMID 26807110
- [Background] Lonskaya I, Hebron ML, Selby ST, Turner RS, Moussa CE. Nilotinib and bosutinib modulate pre-plaque alterations of blood immune markers and neuro-inflammation in Alzheimer's disease models. Neuroscience. 2015 Sep 24;304:316-27. doi: 10.1016/j.neuroscience.2015.07.070. Epub 2015 Jul 30. PMID 26235435
- [Background] Hebron ML, Lonskaya I, Olopade P, Selby ST, Pagan F, Moussa CE. Tyrosine Kinase Inhibition Regulates Early Systemic Immune Changes and Modulates the Neuroimmune Response in alpha-Synucleinopathy. J Clin Cell Immunol. 2014 Sep 30;5:259. doi: 10.4172/2155-9899.1000259. PMID 25635231
- [Background] Lonskaya I, Hebron ML, Desforges NM, Schachter JB, Moussa CE. Nilotinib-induced autophagic changes increase endogenous parkin level and ubiquitination, leading to amyloid clearance. J Mol Med (Berl). 2014 Apr;92(4):373-86. doi: 10.1007/s00109-013-1112-3. Epub 2013 Dec 13. PMID 24337465
- [Background] Hebron ML, Lonskaya I, Moussa CE. Tyrosine kinase inhibition facilitates autophagic SNCA/alpha-synuclein clearance. Autophagy. 2013 Aug;9(8):1249-50. doi: 10.4161/auto.25368. Epub 2013 Jun 19. PMID 23787811
- [Background] Lonskaya I, Hebron ML, Desforges NM, Franjie A, Moussa CE. Tyrosine kinase inhibition increases functional parkin-Beclin-1 interaction and enhances amyloid clearance and cognitive performance. EMBO Mol Med. 2013 Aug;5(8):1247-62. doi: 10.1002/emmm.201302771. Epub 2013 Jul 4. PMID 23737459
- [Background] Folch J, Petrov D, Ettcheto M, Pedros I, Abad S, Beas-Zarate C, Lazarowski A, Marin M, Olloquequi J, Auladell C, Camins A. Masitinib for the treatment of mild to moderate Alzheimer's disease. Expert Rev Neurother. 2015 Jun;15(6):587-96. doi: 10.1586/14737175.2015.1045419. Epub 2015 May 11. PMID 25961655
- [Background] Galvin JE. THE QUICK DEMENTIA RATING SYSTEM (QDRS): A RAPID DEMENTIA STAGING TOOL. Alzheimers Dement (Amst). 2015 Jun 1;1(2):249-259. doi: 10.1016/j.dadm.2015.03.003. PMID 26140284
- [Background] Adamczuk K, Schaeverbeke J, Vanderstichele HM, Lilja J, Nelissen N, Van Laere K, Dupont P, Hilven K, Poesen K, Vandenberghe R. Diagnostic value of cerebrospinal fluid Abeta ratios in preclinical Alzheimer's disease. Alzheimers Res Ther. 2015 Dec 18;7(1):75. doi: 10.1186/s13195-015-0159-5. PMID 26677842
- [Background] Llorens F, Schmitz M, Ferrer I, Zerr I. CSF biomarkers in neurodegenerative and vascular dementias. Prog Neurobiol. 2016 Mar-May;138-140:36-53. doi: 10.1016/j.pneurobio.2016.03.003. Epub 2016 Mar 22. PMID 27016008
- [Background] Teipel SJ, Cavedo E, Grothe MJ, Lista S, Galluzzi S, Colliot O, Chupin M, Bakardjian H, Dormont D, Dubois B, Hampel H; Hippocampus Study Group. Predictors of cognitive decline and treatment response in a clinical trial on suspected prodromal Alzheimer's disease. Neuropharmacology. 2016 Sep;108:128-35. doi: 10.1016/j.neuropharm.2016.02.005. Epub 2016 Feb 10. PMID 26876309
- [Background] Trebeschi S, Riederer I, Preibisch C, Bohn KP, Forster S, Alexopoulos P, Zimmer C, Kirschke JS, Valentinitsch A. Diagnostic Potential of Pulsed Arterial Spin Labeling in Alzheimer's Disease. Front Neurosci. 2016 Apr 19;10:154. doi: 10.3389/fnins.2016.00154. eCollection 2016. PMID 27147946
- [Background] Cortes JE, Kantarjian HM, Brummendorf TH, Kim DW, Turkina AG, Shen ZX, Pasquini R, Khoury HJ, Arkin S, Volkert A, Besson N, Abbas R, Wang J, Leip E, Gambacorti-Passerini C. Safety and efficacy of bosutinib (SKI-606) in chronic phase Philadelphia chromosome-positive chronic myeloid leukemia patients with resistance or intolerance to imatinib. Blood. 2011 Oct 27;118(17):4567-76. doi: 10.1182/blood-2011-05-355594. Epub 2011 Aug 24. PMID 21865346
- [Background] Jefferson AL, Beiser AS, Seshadri S, Wolf PA, Au R. APOE and mild cognitive impairment: the Framingham Heart Study. Age Ageing. 2015 Mar;44(2):307-11. doi: 10.1093/ageing/afu183. Epub 2014 Dec 11. PMID 25497326
- [Background] Janofsky JS, McCarthy RJ, Folstein MF. The Hopkins Competency Assessment Test: a brief method for evaluating patients' capacity to give informed consent. Hosp Community Psychiatry. 1992 Feb;43(2):132-6. doi: 10.1176/ps.43.2.132. PMID 1572608
- [Background] Appelbaum PS. Clinical practice. Assessment of patients' competence to consent to treatment. N Engl J Med. 2007 Nov 1;357(18):1834-40. doi: 10.1056/NEJMcp074045. No abstract available. PMID 17978292